CLINICAL TRIAL: NCT00213850
Title: Reference Values for Respiratory Resistance Measured by the Interrupter Technique in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2667
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Interrupter technique; Respiratory resistance; Normal adults

INTERVENTIONS:
Procedure: EFR

SUMMARY:
The purpose is to obtain reference values of respiratory resistance (a technique widely used in children), in adults. The interest is that this technique needs only little co-operation and would be particularly adapted in subjects in whom co-operation is insufficient for other measurements.

ELIGIBILITY:
Inclusion Criteria:

* Adult non smokers, without any disease interfering with pulmonary function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2002-01; Study Completion 2006-09

PRIMARY OUTCOMES:
References values obtained once

SECONDARY OUTCOMES:
Estimation of short-term reproductibility

CONTACTS AND LOCATIONS:
Overall Officials: Monique OSWALD-MAMMOSSER, MD, Principal Investigator — Service de Physiologie Clinique et des Explorations Fonctionnelles, Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Physiologie Clinique et des Explorations Fonctionnelles, Hôpital Civil, Strasbourg, France

REFERENCES:
- [Result] Oswald-Mammosser M, Charloux A, Enache I, Lonsdorfer-Wolf E. The opening interrupter technique for respiratory resistance measurements in children. Respirology. 2010 Oct;15(7):1104-10. doi: 10.1111/j.1440-1843.2010.01828.x. PMID 20874747